CLINICAL TRIAL: NCT00703898
Title: Durability of Stavudine, Lamivudine and Nevirapine Among Advanced HIV-1 Infected Patients With/Without Prior Co-Administration of Rifampicin: A 144-Week Prospective Study
Brief Title: Durability of Nevirapine-Based Antiretroviral Regimen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bamrasnaradura Infectious Diseases Institute (Other Government)
Responsible Party: Weerawat Manosuthi, Bamrasnaradura Infectious Diseases Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0327/3619
Record Dates: First submitted 2008-06-20; First posted 2008-06-24 (Estimated); Last update posted 2008-07-08 (Estimated); Status verified 2008-06

CONDITIONS: HIV Infections
Keywords: HIV; nevirapine; durability; AIDS; Treatment Naïve
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Nevirapine; stavudine, lamivudine, nevirapine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: nevirapine — 200 mg/day twice a day
  Other Names: GPO-vir

SUMMARY:
Although nevirapine is used as an alternative to efavirenz for initial regimen in developed countries, nevirapine has still been a key antiretroviral drug in many resource-limited countries including Thailand due to its accessibility and affordability. In addition, a component of stavudine and lamivudine is still widely used as a backbone in the antiretroviral regimen in this setting.To date, data on the durability of a regimen of stavudine, lamivudine and nevirapine are very limited, particularly from the resource-limited settings.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected individuals ≥15 years of age
* CD4 cell count <350 cells/mm3
* Willing to participate and give consent form

Exclusion Criteria:

* previous antiretroviral therapy
* pregnancy
* receiving a medication that has drug-drug interactions with NVP or RFP
* aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >5 times of upper limit of normal range

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2004-11; Primary Completion 2009-12; Study Completion 2010-04

PRIMARY OUTCOMES:
number of patients with undetectable plasma HIV-1 viral load | 240 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Weerawat Manosuthi, Principal Investigator — Bamrasnaradura Infectious Diseases Institute
Locations (1):
- Department of Medicine, Bamrasnaradura Infectious Diseases Institute, Nonthaburi, Changwat Nonthaburi, Thailand

REFERENCES:
- [Derived] Manosuthi W, Tantanathip P, Prasithisirikul W, Likanonsakul S, Sungkanuparph S. Durability of stavudine, lamivudine and nevirapine among advanced HIV-1 infected patients with/without prior co-administration of rifampicin: a 144-week prospective study. BMC Infect Dis. 2008 Oct 14;8:136. doi: 10.1186/1471-2334-8-136. PMID 18851761